CLINICAL TRIAL: NCT00944801
Title: RNOP-09: Pegylated Liposomal Doxorubicine and Prolonged Temozolomide in Addition to Radiotherapy in Newly Diagnosed Glioblastoma - a Phase II Study
Brief Title: Pegylated Liposomal Doxorubicine and Prolonged Temozolomide in Addition to Radiotherapy in Newly Diagnosed Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: Essex Pharma Germany (Other)
Responsible Party: Ulrich Bogdahn, Prof. Dr. med., Department of Neurology, University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNOP-09
Record Dates: First submitted 2009-07-17; First posted 2009-07-23 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Glioblastoma
Keywords: glioblastoma; first-line; clinical trial; PEG-liposomal doxorubicin; temozolomide; radiotherapy; phase 1; phase 2
MeSH Terms: conditions — Glioblastoma | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pegylated Liposomal Doxorubicin (Experimental): Radiotherapy is planned with dedicated computed tomography and three-dimensional planning systems and delivered to the gross tumor volume with a 2 to 3 cm margin for the clinical target volume. After a 4-week break, patients receive adjuvant TMZ 150 to 200 mg/m2 day 1 to 5 in 28 days until tumor progression or up to at least 12 cycles. In the dose escalation phase of the study, PEG-Dox is raised in steps of 5 mg/m2 in a 3-by-3 design, starting with 5 mg/m2 (group 1) up to 20 mg/m2 (group 4). In the phase II part of the study, the targeted dose of 20 mg/m2 is administered up to a cumulative dose of 550 mg/m2 or until tumor progression.
  Interventions: Drug: Pegylated Liposomal Doxorubicine

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicine — In the dose escalation phase of the study, PEG-Dox is raised in steps of 5 mg/m2 in a 3-by-3 design, starting with 5 mg/m2 (group 1) up to 20 mg/m2 (group 4). In the phase II part of the study, the targeted dose of 20 mg/m2 is administered up to a cumulative dose of 550 mg/m2 or until tumor progression.
  Other Names: Caelyx

SUMMARY:
Glioblastomas represent 40% of all tumors of the central nervous system (CNS) and are among the most lethal tumors. Temozolomide (TMZ) combined with radiotherapy was the first substance to significantly improve the overall survival (to 14.6 months) as compared to surgery and radiotherapy alone and increased the proportion of patients surviving more than 2 years to 26%. TMZ showed the best efficacy in patients with a methylated O6-methylguanine-DNA methyltransferase (MGMT) promoter in part by eliminating stem cell-like tumor cells. Among patients with a methylated MGMT promoter, the median survival after treatment with combined radio-chemotherapy was 21.7 months, as compared to 15.3 months among those who were assigned to radiotherapy only. In the absence of methylation of the MGMT promoter, there was a smaller and statistically insignificant difference in survival between the treatment groups.

Doxorubicin is one of the most effective substances in vitro against cells derived from glioblastoma. However, it has no significant effect in vivo due to poor blood-brain-barrier penetration. In a tumor model, tissue and CSF-concentrations of doxorubicin were substantially increased when sterically stabilized liposomes were used resulting in a comparable clinical response using approximately half of the dose of stabilized liposomes compared to conventional doxorubicin. A pegylated formulation (PEG-liposomal Doxorubicin) even further improved the penetration of the blood-brain barrier. Case series and two phase II-studies in patients with recurrent glioblastoma have shown modestly promising results for PEG-Dox.

In this study, the investigators treated patients with recurrent glioblastoma with 20 mg/m2 PEG-Dox on days 1 and 15 of each 28-day cycle. To determine the dose limiting toxicity of PEG-Dox combined with prolonged administration of TMZ, the investigators performed a phase I part ahead of the phase II study. To investigate, by means of a historical control analysis, if the addition of PEG-Dox to TMZ and radiotherapy improves the survival of patients, the investigators chose similar inclusion criteria and identical TMZ and radiotherapeutic regimes as in the EORTC26981/NCIC-CE.3 study.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed glioblastoma
* centrally confirmed histology
* Karnofsky performance score (KPS) > 70%
* stable corticosteroids within 2 weeks before inclusion
* leucocytes > 3/ul, thrombocytes > 100/ul, Hb > 10 g/dl
* additional standard criteria

Exclusion Criteria:

* other tumor in history
* pretreatment with radiotherapy to the brain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2002-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
progression free survival probability at 12 months to detect an improvement of the PFS-12 of 15.6% as compared to EORTC26981/NCIC-CE.3 combination arm (PFS-12: 26.9%) | 12 months after inclusion of last patient

SECONDARY OUTCOMES:
PFS-24, mOS, OS-12, OS-24, mTTP, response rate, rate of stabilizations , and toxicity profile | 12 months after inclusion of last patient

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Bogdahn, MD, Prof., Principal Investigator — Department of Neurology, University of Regensburg
Locations (1):
- University of Regensburg, Department of Neurology, Regensburg, Germany

REFERENCES:
- [Derived] Beier CP, Schmid C, Gorlia T, Kleinletzenberger C, Beier D, Grauer O, Steinbrecher A, Hirschmann B, Brawanski A, Dietmaier C, Jauch-Worley T, Kolbl O, Pietsch T, Proescholdt M, Rummele P, Muigg A, Stockhammer G, Hegi M, Bogdahn U, Hau P. RNOP-09: pegylated liposomal doxorubicine and prolonged temozolomide in addition to radiotherapy in newly diagnosed glioblastoma--a phase II study. BMC Cancer. 2009 Sep 2;9:308. doi: 10.1186/1471-2407-9-308. PMID 19725960